CLINICAL TRIAL: NCT06793358
Title: Use of Remimazolam and Fentanyl for Procedural Sedation in Patients Undergoing Dental Extraction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Kyle J. Kramer, DDS, MS, Clinical Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22891
Record Dates: First submitted 2024-12-16; First posted 2025-01-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Dental Extraction
Keywords: Extraction; sedation; fentanyl; Remimazolam; dental
MeSH Terms: interventions — Fentanyl; remimazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fentanyl and Remimazolam combined (Experimental): Remimazolam has received FDA approval for procedural sedation in adults undergoing procedures lasting 30 minutes or less. While remimazolam has been used in studies for procedural sedation outside of dentistry and oral surgery, there are no dental studies from the US that have assessed its safe and effect use along with fentanyl as described in the package insert. This single-armed study will assess the efficacy of FDA-approved remimazolam combined with fentanyl for procedural sedation (defined as MOAA/S score ≥2) in healthy (ASA 1 and 2) adults undergoing dental extractions expected to last 30 minutes or less. To date, there are no studies in the US that have assessed the effectiveness of remimazolam and fentanyl for procedural sedation for dental treatment, including extractions, so this is the first study of its kind.
  Interventions: Drug: fentanyl and Remimazolam

INTERVENTIONS:
Drug: fentanyl and Remimazolam — This is the first dental study that will combine these two sedation drugs

SUMMARY:
The goal of this clinical trial is to learn if a combination of the two established sedation drugs remimazolam and fentanyl, can put the subject to sleep during a scheduled extraction procedure. The combined use of these drugs has been used in other studies involving IV sedation when the procedure is scheduled for 30 minutes or less. However, the combined use of the IV sedation drugs has not been used in a dental extraction procedure before.

The main questions it aims to answer are:

1. Can the combined drugs effectively put the patient to sleep during the procedure
2. How quickly will they come out of the sedation after the procedure

Participants will:

1. Receive the combined drugs during a scheduled extraction procedure anticipated to take less than 30 minutes
2. Answer survey questions related to their study experience after the extraction visit (in person) and again about 24 hours after the visit (by telephone).

DETAILED DESCRIPTION:
Primary Objective The Primary objective of this study is to determine if the combination of remimazolam and fentanyl for IV procedural sedation is effective for completion of the planned surgical procedure (a composite of MOAA/S scores of 2-4, extraction of indicated teeth, no need for rescue medications [propofol, flumazenil]).

Secondary Objective Secondary objectives include determination of the speed of emergence and recovery from sedation as calculated by the total anesthesia time, total surgery time, time from end of surgery to emergence and fitness for discharge (modified Aldrete score ≥9, minimal/no PONV, pain controlled).

Tertiary/Exploratory/Correlative Objectives Other measured data will include changes in blood pressure and heart rate (+/- 20% of baseline); emergent/urgent use of vasoactive agents; changes in ventilation/oxygenation (hypoxemia, SpO2 <90%; rescue ventilation), MOAA/S scores <2, and other rare sedation complications (PONV, anaphylaxis, etc.).

Study Design This will be a single arm, single site, unblinded clinical trial using two marketed intravenous sedation drugs (remimazolam and fentanyl) to determine whether this drug combination is effective for dental extractions under procedural sedation.

Neither the study team member administering the study drugs, nor the participant will be blinded to the sedation drug they are receiving. Blinding is not necessary at this time since the study is a single-arm design.

Written informed consent will be obtained prior to any study procedures being performed.

Enrollment/Randomization Potential subjects will be patients who are scheduled for dental extractions under sedation in the IUSD Oral Surgery Clinic at IU Health University Hospital. Recruitment will occur chairside during the consultation appointment or at the extraction appointment, and up to 40 participants will receive remimazolam and fentanyl for procedural sedation as the IV sedatives for their planned dental extractions.

Study Procedures

Following the consenting procedure, the following will be performed:

1. The patient will be weighed preoperatively (recorded in kg) and confirmation of adherence to NPO instructions (nothing by mouth) and presence of an escort will occur as per usual. The patient will then be escorted and seated in the dental operatory.
2. Inclusion/Exclusion criteria will be reviewed to confirm eligibility.
3. A dental exam and review of radiographs, collected as standard of care, will be performed along with confirmation of planned extractions.
4. Preparation of the study drugs will occur in the standard, sterile fashion.
5. Upon arrival to the dental operatory, standard anesthesia monitors (ECG, pulse oximetry, noninvasive BP cuff, nasal capnography, precordial stethoscope) will be placed. Supplemental oxygen at 4 L/min will be supplied via nasal cannula with CO2- carbon dioxide (capnography) monitoring capabilities.
6. Preoperative vital signs (BP, HR (heart rate), RR (respiratory rate), room air SpO2) will be obtained after which an IV catheter will be placed in a suitable hand or antecubital vein in order to administer IV fluids (normal saline) and medications. Timing of the successful IV catheter placement will be recorded (anesthesia start time)
7. Study drugs will be administered by a qualified study team member with notation of the time study drug administration began documented along with the dose.
8. Study drug dosing will follow the same dosing protocol as documented in the initial Phase 3 trials. IV boluses of remimazolam (5 mg initially/2.5 mg additional boluses ≥2 min apart) and fentanyl (25-50 mcg initially/25 mcg additional boluses every 5-10 minutes; up to 100 mcg total) will be administered and titrated to desired procedural sedation level (MOAA/S: 2-4).
9. Upon confirming targeted sedation depth has been achieved, the vital signs will be reassessed. A rubber bite block will then be placed intraorally, and the operating surgeon will administer local anesthetic solution (2% lidocaine with 1:100,000 epinephrine) as per usual. Local anesthetic total volumes will be documented along with the technique. Local anesthetics used are standard of care in any extraction procedure.
10. Vital signs will be re-assessed 3 minutes after completing the local anesthetic injections and re-assessed every 5 minutes thereafter.
11. The dental extractions will then be completed as per the departmental standard of care. Time of commencement of the extractions (surgery start time) will be recorded. The procedure will be observed by a study team member who will document any unusual occurrences that might be related to the study drug.
12. Time of completion of the extractions (surgery end time) will be recorded as well as the time of the last dose of either study drug (remimazolam or fentanyl).
13. Patient will be gently shaken and asked to open their eyes immediately after surgery stop. This will be repeated every 1 minute until patient is able to comply. Time of eye opening will be recorded.
14. Patient will remain seated and monitored until assessed and determined that they are fit for discharge. Assessment will occur every minute, and this time will be recorded (anesthesia stop). Fitness for discharge will include modified Aldrete score ≥9, controlled pain, minimal/no PONV).
15. If needed for rescue due to failed/insufficient sedation, or if the procedure extends beyond the 30 minute allowance for the study drugs, propofol and/or midazolam will be used to facilitate safe completion of the planned surgical procedure as per usual. Ondansetron (0.1 mg/kg up to 4 mg total) will be used for PONV rescue if the patient experiences nausea and/or vomiting postoperatively prior to discharge as per usual. All drugs listed here are considered standard of care for dental sedation procedures. If rescue drugs are administered, the use of the rescue drug will be documented in the study procedures. The subjects will be withdrawn from the study at the point of rescue drug administration and no additional study procedures will be followed or recorded from this point forward.
16. Prior to discharge home, the patient will be asked to complete the Patient Satisfaction Survey which consists of 5 questions answered using a 5-point Likert scale. This survey will be repeated within 24 hours on postoperative day 1 via telephone.
17. The operating surgeon will complete a satisfaction survey using a 5-point Likert scale after the procedure is complete.
18. Patients will be asked to follow up with their operating surgeon at the same clinic as per usual. Instructions will be given to the patient and escort prior to discharge detailing contact information in case any adverse events/reactions occur afterwards per usual. All other postoperative instructions and analgesic prescriptions will follow established departmental standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Willing to read and sign the IRB (Institutional Review Board) approved informed consent document.
* Patients 18 years of age and older on the day of the surgery
* Healthy patients (ASA Physical Status class of 1 or 2)
* Dental treatment consists of planned extractions expected to be completed in 30 minutes or less using IV moderate (procedural) sedation.

Exclusion Criteria:

List the criteria:

* Allergy or negative history with either of the planned sedative medications (remimazolam, fentanyl) or local anesthetics to be used for dental extractions.
* Previous negative history with the use of IV sedation medications
* Use of opioid-containing analgesics within 24 hours of surgery
* BMI >30 kg/m2
* Patients with multiple or poorly controlled medical comorbidities (i.e., hypertension, COPD (chronic obstructive pulmonary disease), heart failure, asthma, diabetes).
* Consumption within the last 24 hours of alcohol, illicit (marijuana, cocaine, etc.), opioid-containing, or other analgesic drugs.
* Other contraindications to procedural/moderate sedation (i.e., concurrent illness, failure to follow NPO (nil per os) instructions, lack of escort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure for IV Sedation for completion of Surgery using successful extraction of teeth (1) | 30 minutes extraction period at the end of surgery
  Successful extraction of the indicated teeth (assessed at end of surgery)
Primary Outcome Measure for IV Sedation for completion of Surgery (2) using MOAA/s scores ( | 30 minutes extraction period at the end of surgery
  Maximum MOAA/S scores (Modified Observer's Assessment of Alertness and Sedation Score) of 2-4 during the procedure (score rande of 0 to 6 with 0 meaning no response to stimulus (assessed every 5 minutes)
Primary Outcome Measure for IV Sedation for completion of Surgery determined by no need for rescue medications (3) | 30 minutes extraction period at the end of surgery
  No need for rescue medications (propofol, flumazenil, naloxone).

SECONDARY OUTCOMES:
Secondary Outcome Measure related to timing related to anesthesia length, surgery, eye opening and discharge | 30 minutes extraction period at the end of surgery
  Time associated with anesthesia length, surgery length,eye opening, discharge

OTHER OUTCOMES:
Other measured data related to sedation depth (1) | 30 minutes extraction period at the end of surgery
  Sedation depth greater than intended (MOAA/S scores <2)
Other measured data related to other rare sedation complications (2) | 30 minutes extraction period at the end of surgery
  Assessing for other rare sedation complications (PONV, anaphylaxis, etc)
Blood pressure during extraction period | Every 5 minutes throughout the 30 minute extraction period
  Blood pressure every 5 minutes
Heart rate during extraction period | Every 5 minutes throughout the 30 minute extraction period
  Heart rate every 5 minutes
Other measured data related to emergent/urgent use of vasoactive agents(4) | 30 minutes extraction period at the end of surgery
  Emergent/urgent use of vasoactive agents (i.e, atropine, ephedrine, phenylephrine, epinephrine, etc.)
Other measured data Hypoxemia (5) | 30 minutes extraction period at the end of surgery
  Hypoxemia (SpO2 <90%), need for rescue ventilation,
Other measured data total drug doses for all drugs administered in the study (6) | 30 minutes extraction period at the end of surgery
  Total drug doses for all drugs administered in the study (remimazolam, fentanyl, local anesthetics, rescue/emergency drugs)

CONTACTS AND LOCATIONS:
Overall Officials: kyle j kramer, DDS, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Dentistry (IUSD), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided